CLINICAL TRIAL: NCT04995055
Title: Evaluation of Multifocal Contact Lens Designs With and Without an HEV Blocker on Visual Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-6391
Record Dates: First submitted 2021-07-29; First posted 2021-08-06 (Actual); Results first posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Period 1 (Experimental): Eligible subjects will be randomly assigned to contact lens wear sequence TEST/CONTROL in a bilateral fashion.
  Interventions: Device: JJVC Investigational Multifocal Contact Lens TEST Lens; Device: ACUVUE® OASYS Multifocal
- Period 2 (Experimental): Eligible subjects will be randomly assigned to contact lens wear sequence CONTROL/ TEST in a bilateral fashion.
  Interventions: Device: JJVC Investigational Multifocal Contact Lens TEST Lens; Device: ACUVUE® OASYS Multifocal

INTERVENTIONS:
Device: JJVC Investigational Multifocal Contact Lens TEST Lens — TEST Lens
Device: ACUVUE® OASYS Multifocal — CONTROL Lens

SUMMARY:
This is a single-masked, bilateral, controlled, randomized, 2x2 crossover, non-dispensing clinical trial to characterize the effects of an HEV-Blocker on several measures of visual function in a presbyopic population.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

  1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form
  2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. Be between at least 40 and not more than 70 years of age at the time of screening.
  4. Possess a wearable pair of spectacles that provide correction for distance vision.
  5. Be an adapted soft contact lens wearer in both eyes (i.e. worn lenses a minimum of 2 days per week for at least 8 hours per wear day, for 1 month of more duration).
  6. Be wearing a presbyopic contact lens correction (e.g., reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or if not respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire".
  7. The subject must have normal color perception as evidenced by reading 17 out of the first 21 Ishihara plates correctly.
  8. The subject's distance spherical equivalent of their refraction must be in the range of -1.00 D to -4.00 D.
  9. The subject's refractive cylinder must be ≤0.75 D in each eye.
  10. The subject's ADD power must be in the range of +0.75 D to +2.50 D in each eye.
  11. The subject must have best corrected distance visual acuity of 20/20-3 or better in each eye.

      Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Be currently pregnant or lactating.
  2. Any systemic disease (e.g., Sjögren's Syndrome), allergies, infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive diseases (e.g., HIV), autoimmune disease (e.g. rheumatoid arthritis), or other diseases, by self-report, which are known to interfere with contact lens wear and/or participation in the study.
  3. Use of any of the following oral medications within 1 week prior to enrollment: oral retinoids, oral tetracyclines, oral phenothiazines, anticholinergics, oral/inhaled steroids, oral phosphodiesterase type 5 inhibitors, interferon alfa, antimycobacterial antibiotics, and nitroimidazole antibiotics. See Section 9.1 for additional details regarding excluded systemic medications.
  4. Any current use of ocular medication with the exception of rewetting drops.
  5. Any known hypersensitivity or allergic reaction to single use preservative free rewetting drops or sodium fluorescein.
  6. Any previous or planned (during the course of the study) ocular surgery (e.g., radial keratotomy, PRK, LASIK dacryocystorhinostomy, cataract surgery, retinal surgery, peripheral iridotomy/iridectomy, etc.).
  7. Participation in any contact lens or lens care product clinical trial within 7 days prior to study enrollment.
  8. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
  9. Any active or ongoing ocular or systemic allergies that may interfere with contact lens wear.
  10. A history of amblyopia, strabismus or binocular vision abnormality.
  11. History of optic nerve or retinal disease or trauma
  12. Abnormal color vison.
  13. Any other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, or corneal distortion
  14. Any grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA scale.
  15. Any current ocular infection or inflammation.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (1):
- University of Georgia, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 37 subjects were enrolled into this study. Of those enrolled, 35 were fit into at least 1 study lens, while 2 subjects failed to meet all eligibility criteria. Of those dispensed, 25 subjects completed the study, while 10 subjects were discontinued.
Groups:
- Senofilcon A\Senofilcon A (C3): Subjects randomized to this sequence received the senofilcon A lens during the first period and then received the senofilcon A (C3) lens during the second period
- Senofilcon A (C3)\ Senofilcon A: Subjects randomized to this sequence received the senofilcon A (C3) lens during the first period and then received the senofilcon A lens during the second period
Period: Period 1
Arm/Group | Senofilcon A\Senofilcon A (C3) | Senofilcon A (C3)\ Senofilcon A
Started | 17 | 18
Completed | 12 | 13
Not Completed | 5 | 5
Not completed — COVID-19 Related | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Subject discontinued due to timing | 4 | 4
Period: Period 2
Arm/Group | Senofilcon A\Senofilcon A (C3) | Senofilcon A (C3)\ Senofilcon A
Started | 12 | 13
Completed | 12 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects fitted at least one study lens.
Groups:
- Fitted Subjects: All subjects fitted at least one study lens.
Arm/Group | Fitted Subjects
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.8 (7.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 5
Race/Ethnicity, Customized [Number; unit: Participants]
  Black or African American | 6
  White | 29
Region of Enrollment [Number; unit: Participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Starburst Diameter (mm)
Description: The starburst diameter (mm) was measured each subject binocularly. Starburst diameter was quantified by the horizontal spread of the spokes emerging from the center of a small, point-like stimulus. A calibrated custom-made micrometer (two sides with reverse threading) was used to spread two posts out from a central mid-point. The posts attach to a custom-designed ruler that indicates the lateral spread of the starburst. Measurements for this metric are positive. Smaller diameter indicates better lens performance. The average diameter (mm) for each lens type was reported by period.
Time Frame: 30-minutes post lens insertion
Population: All subjects fitted at least one study lens.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Senofilcon A: Subjects that wore senofilcon A lens in either the first or second period of the study.
- Senofilcon A (C3): Subjects that wore senofilcon A (C3) lens in either the first or second period of the study.
Arm/Group | Senofilcon A | Senofilcon A (C3)
Number analyzed (Participants) | 30 | 30
mm
  Period 1: number analyzed (Participants) | 17 | 18
  Period 1 | 77.06 (25.900) | 64.13 (27.703)
  Period 2: number analyzed (Participants) | 13 | 12
  Period 2 | 67.26 (30.991) | 54.24 (22.706)

2. Primary Outcome: Halos Diameter (mm)
Description: Halo diameter (mm) was quantified and measured using the same micrometer as for starbursts diameter (mm). The Halo diameter (mm) was measured each subject binocularly. Measurements for halo diameter are positive, where smaller values indicate better performance. The average diameter (mm) for each lens type.
Time Frame: 30-minutes post lens insertion
Population: All subjects fitted at least one study lens.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Senofilcon A | Senofilcon A (C3)
Number analyzed (Participants) | 30 | 30
mm | 69.24 (19.033) | 52.93 (17.725)
Statistical Analysis 1: Comparison: Senofilcon A vs Senofilcon A (C3); Test type: Superiority; Linear Mixed Model; Kenward and Roger method was used for denominator degrees of freedom; Least-square Mean Difference = -15.4, 95% CI 2-sided [-21.2 to -9.5], Standard Error of Mean 2.81 — Least-square Mean difference was calculated as senofilcon A (C3)- senofilcon A

3. Primary Outcome: Glare Disability Threshold
Description: Glare disability threshold was collected binocularly for each subject. Subjects were exposed to a target stimulus for 2 seconds; before the measurement was taken the annulus was set to a level below that which would cause the target stimulus to be veiled. The experimenter would then adjust the intensity of the annulus until subjects could no longer see the target stimulus. Subjects would indicate this by pressing a buzzer. Glare disability thresholds take on positive values, where higher values indicate better lens performance. The average glare disability level (change in log relative energy) for each lens type was reported.
Time Frame: 30-minutes post lens insertion
Population: All subjects fitted at least one study lens.
Measure: Mean (Standard Deviation); unit: log (change in log relative energy)
Arm/Group | Senofilcon A | Senofilcon A (C3)
Number analyzed (Participants) | 30 | 29
log (change in log relative energy) | 2.62 (0.235) | 2.86 (0.179)
Statistical Analysis 1: Comparison: Senofilcon A vs Senofilcon A (C3); Test type: Superiority; Linear Mixed Model; Kenward and Roger method was used for denominator degrees of freedom; Least-square Mean Difference = 0.3, 95% CI 2-sided [0.2 to 0.4], Standard Error of Mean 0.04 — Least-square Mean difference was calculated as senofilcon A (C3)- senofilcon A

4. Secondary Outcome: Glare Discomfort (mm)
Description: The Glare discomfort was evaluated by calculating the change in height of the palpebral fissure measured while the participant views the mid-wave central grating target, compared to the maximal squint during a 5-second Photostress exposure induced by a solid, 10-degree broadband field, which completely obscures the target (~10-deg diameter). Both eyes were recorded and averaged, to produce an average palpebral fissure height before and during the Photostress exposure. Glare discomfort can take on negative and positive values, where smaller values indicate better lens performance. The average glare discomfort (change in palpebral fissure height) for each lens type was reported.
Time Frame: 30-minutes post lens insertion
Population: All subjects fitted at least one study lens.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Senofilcon A | Senofilcon A (C3)
Number analyzed (Participants) | 30 | 30
mm | 9.88 (4.164) | 6.61 (3.151)
Statistical Analysis 1: Comparison: Senofilcon A vs Senofilcon A (C3); Test type: Superiority; Linear Mixed Model; Kenward and Roger method was used for denominator degrees of freedom; Least-square Mean Difference = -3.5, 95% CI 2-sided [-4.9 to -2.1], Standard Error of Mean 0.66 — Least-square Mean difference was calculated as senofilcon A (C3)- senofilcon A

5. Secondary Outcome: Heterochromatic Contrast Threshold (HCT)
Description: Using the same optical bench set-up described Glare Disability Threshold, to measure HCT, participants viewed the mid-wave (580 nm) grating target presented on presented on a short wave (460 nm) "sky-light background." The intensity of the background was adjusted, until the participant was no longer able to resolve the grating target. The log relative energy of the background needed to obscure the central target was recorded as HCT. Heterochromatic contrast thresholds are positive values, where higher values indicate better lens performance. The average threshold each lens type was reported.
Time Frame: 30-minutes post lens insertion
Population: All subjects fitted at least one study lens.
Measure: Mean (Standard Deviation); unit: log (change in log relative energy)
Arm/Group | Senofilcon A | Senofilcon A (C3)
Number analyzed (Participants) | 30 | 29
log (change in log relative energy) | 1.85 (0.221) | 2.14 (0.295)
Statistical Analysis 1: Comparison: Senofilcon A vs Senofilcon A (C3); Test type: Superiority; Linear Mixed Model; Kenward and Roger method was used for denominator degrees of freedom; Least-square Mean Difference = 0.3, 95% CI 2-sided [0.2 to 0.4], Standard Error of Mean 0.05 — Least-square Mean difference was calculated as senofilcon A (C3)- senofilcon A

6. Secondary Outcome: Two-Point Threshold (mm) With 403nm Filter
Description: To create the two-point threshold stimulus, a single point- source like stimulus was spread into two distinct points of light, using a custom-built, collapsible light baffle. The two-point threshold was quantified as the minimum distance (mm) at which a participant could detect two distinct points of light, separated by a small black space. Measurements for this metric are positive. Smaller distances indicate better lens performance. The average distance for each lens type and period.
Time Frame: 30-minutes post lens insertion
Population: All subjects fitted at least one study lens.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Senofilcon A | Senofilcon A (C3)
Number analyzed (Participants) | 30 | 30
mm
  Period 1: number analyzed (Participants) | 17 | 18
  Period 1 | 16.49 (5.600) | 7.51 (2.889)
  Period 2: number analyzed (Participants) | 13 | 12
  Period 2 | 13.21 (5.021) | 9.50 (6.321)

7. Secondary Outcome: Two-Point Threshold (mm) Without 403nm Filter
Description: To create the two-point threshold stimulus, a single point- source like stimulus was spread into two distinct points of light, using a custom-built, collapsible light baffle. The two-point threshold was quantified as the minimum distance (mm) at which a participant could detect two distinct points of light, separated by a small black space. Measurements for this metric are positive. Smaller distances indicate better lens performance. The average distance for each lens type.
Time Frame: 30-minutes post lens insertion
Population: All subjects fitted at least one study lens.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Senofilcon A | Senofilcon A (C3)
Number analyzed (Participants) | 30 | 30
mm | 8.63 (3.391) | 5.47 (1.953)
Statistical Analysis 1: Comparison: Senofilcon A vs Senofilcon A (C3); Test type: Superiority; Linear Mixed Model; Kenward and Roger method was used for denominator degrees of freedom; Least-square Mean Difference = -3.1, 95% CI 2-sided [-4.4 to -1.9], Standard Error of Mean 0.59 — Least-square Mean difference was calculated as senofilcon A (C3)- senofilcon A

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study; approximately 5- 10 days per subject.
Groups:
- Senofilcon A: Subjects that wore the senofilcon A lens during either period of the study.
Arm/Group | Senofilcon A (C3) | Senofilcon A
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-12): https://cdn.clinicaltrials.gov/large-docs/55/NCT04995055/Prot_SAP_000.pdf